CLINICAL TRIAL: NCT05033626
Title: Simultaneous Operations on the Thyroid Gland and Hyoid Suspension in Patients With Combined Thyroid Pathology and Obstructive Sleep Apnea (OSA).
Brief Title: Simultaneous Operations on the Thyroid Gland and Hyoid Suspension in Patients With Combined Thyroid Pathology and OSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Principal Investigator, Oleg Savchuk, Associated professor, Principal Investigator, State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMSC-02-21
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea; Obstructive Sleep Apnea-hypopnea; Obstructive Sleep Apnea-hypopnea Syndrome
Keywords: OSA, CPAP, hyoid suspension, hypopharyngeal obstruction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Microcephaly, Primary Autosomal Recessive, 6 | interventions — Thyroidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyroidectomy (Other)
  Interventions: Procedure: Thyroidectomy
- Simultaneous thyroidectomy and hyoid suspension (Experimental)
  Interventions: Procedure: Simultaneous thyroidectomy and hyoid suspension; Procedure: Thyroidectomy

INTERVENTIONS:
Procedure: Simultaneous thyroidectomy and hyoid suspension — Under endotracheal anesthesia, a horizontal skin incision up to 50 mm long is made at the level of the upper thyroid cartilage, the skin and subcutaneous fat are dissected. The sternohyoid and sternothyroid muscles are retracted. An audit of the thyroid gland is performed. Step by step, using the ultrasonic dissector, the sections of the gland necessary for resection are separated, ligated and transected. Using microsurgical techniques, neurolysis of the recurrent laryngeal nerves is performed. The quality control of the return of the laryngeal nerves is ensured to the required extent using the neuromonitoring apparatus.
  Arms: Simultaneous thyroidectomy and hyoid suspension
Procedure: Thyroidectomy — The hyoid bone is mobilized in the anterocaudal direction and is fixed to the thyroid cartilage with four permanent non-absorbable sutures. If sufficient mobilization does not occur during the operation, the tendon of the stylohyoid muscle is dissected. Surgical drainage is installed 24 hours after surgery.

SUMMARY:
Simultaneous operations on the thyroid gland and hyoid suspension in patients with combined thyroid pathology and moderate to severe OSA.

DETAILED DESCRIPTION:
The ineffectiveness of conservative treatment of obstructive sleep apnea syndrome (OSAS) (CPAP-therapy) or its rejection leads to a surgical solution of the issue, the purpose of which is to eliminate obvious anatomical obstacles, to increase the lumen of the upper respiratory tract. Modern methods of multilevel surgical treatment of OSAS make it possible to achieve more than 80% success.

Most often, at the first stage of OSAS treatment, otorhinolaryngologists use rhinosurgical techniques such as septoplasty, lower submucosal vasotomy, partial conchotomy, removal of nasal polyps, including using endoscopic techniques. At the subsequent stages of multilevel treatment, depending on the level of obstruction and the severity of OSAS, uvulopalatoplasty or uvulopalatopharyngoplasty, partial resection of the tongue or lingual tonsil, suspension of the tongue root and sublingual system, various types of genioplasty and maxillary reduction are performed.

This approach allows expanding the airways in the oropharyngeal region and laryngopharynx, improving functional outcomes and quality of life in patients with OSAS.

At the same time, first of all, it is necessary to carefully assess the benefits and potential risks of surgical treatment, especially in patients with an unfavorable morbid background and from older age groups.

• The investigators will offer patients with concomitant thyroid pathology and moderate or severe OSAS to perform simultaneous operations from one access, where the hyoid bone to the thyroid cartilage will be sutured in the second stage. The stabilization of the hyoid bone and the muscular frame, as an integral complex of the laryngopharynx, increases the airway space and neutralizes obstruction. (1-3) Under endotracheal anesthesia, a horizontal skin incision up to 5 cm long is made at the level of the upper edge of the thyroid cartilage, the skin and subcutaneous fat are dissected. The sternohyoid and sternothyroid muscles are retracted. An audit of the thyroid gland is performed. Step by step, using the ultrasonic dissector, the sections of the gland necessary for resection are separated, ligated, and transected. The vessels of the upper and lower poles are separated with the preservation of blood supply to the right and left upper and lower parathyroid glands. Using a microsurgical technique, neurolysis of the recurrent laryngeal nerves is performed. The control of the integrity of the recurrent laryngeal nerves was performed using the neuromonitoring apparatus.

The hyoid bone is mobilized in the anterocaudal direction and is fixed to the thyroid cartilage with four permanent non-absorbable sutures. If sufficient mobilization does not occur during the operation, the tendon of the stylohyoid muscle is dissected. Surgical drainage is installed 24 hours after surgery.

Advantages:

* access from one incision with combined pathology of the thyroid gland and OSAS which reduces the need for delayed operations;
* decrease in apnea hypopnea index (AHI) to 50.7% and subjective daytime sleepiness according to foreign literature.

ELIGIBILITY:
Inclusion Criteria:

* The patient understands the essence of all procedures planned in the framework of an initiative clinical trial and voluntarily confirms his desire to participate by written informed consent;
* Male or female patients with completed skeletal growth at the age of 30 to 60 years, inclusively, with thyroid pathology and moderate to severe OSAS according to cardiorespiratory monitoring with obstruction of the soft tissues of the upper respiratory tract at the levels of the oropharyngeal and laryngopharynx, without radiography of the pathology of the paranasal sinuses;
* Еhe patient is scheduled for thyroid gland surgery (thyroidectomy with / without lymphadenectomy, subtotal resection of the thyroid gland, hemithyroidectomy).

Exclusion Criteria:

* Women during pregnancy, childbirth;
* Women during breastfeeding;
* Persons with mental disorders;
* Persons detained, taken into custody, serving a sentence in the form of restriction of freedom, arrest, imprisonment or administrative arrest;
* Chronic somatic diseases in the stage of decompensation. Conditions and concomitant pathology of other organs, which are a contraindication for general anesthesia and intubation;
* Diseases and conditions associated with severe bleeding disorders (hemophilia, von Willebrand disease, deficiency of one or more coagulation factors, etc.);
* Infectious diseases in the acute stage.
* Severe brain injuries, which entailed consequences in the form of focal epilepsy, encephalopathy, dementia;
* Pathology of the paranasal sinuses according to X-ray data;
* Pathologies that are relative contraindications for CPAP therapy (bullous lung disease; pulmonary emphysema; a history of pneumothorax, pneumomediastinum, pneumocephalus, respiratory distress syndrome, external liquorrhea; previous surgical interventions on the brain, middle or inner ear, pituitary gland; recurrent sinusitis; recurrent eye infections; severe hypotension; severe dehydration; frequent nosebleeds; fractures of the bones of the face; condition after esophagectomy in history (risk of damage to the anastomosis due to increased pharyngeal / esophageal pressure); hemodynamic instability; a history of severe chronic heart failure; Decompensation of major diseases; cardiomyopathy of any genesis; oncological diseases (except for pathology of the thyroid gland);
* Pathologies that are absolute contraindications for CPAP therapy (unconsciousness of the patient; severe respiratory failure, which may require intubation and subsequent mechanical ventilation; cerebrospinal fluid fistula; collapse of the epiglottis according to sleep endoscopy);
* refusal of the patient to carry out CPAP therapy.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
The absence of severe adverse reactions | Up to 2 months after surgery
  Shortness of breath, bleeding, suppuration

SECONDARY OUTCOMES:
The STOP-BANG questionnaire | Screening, Day 30 and Day 60
  The STOP-BANG questionnaire provides 8 possible signs of the presence of apnea: loud snoring; stopping breathing during sleep; daytime tiredness; increased blood pressure; BMI> 35; neck circumference ≥ 43 cm (41 cm for women), male and over 50 years of age. If there are 3 or more signs, the risk of sleep apnea is considered to be increased.
Three-level European quality of life five-dimensional questionnaire | Screening, Day 30 and Day 60
  There are five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. Patients choice results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describe the health status.
Apnea-Hypopnea Index (AHI) | Screening, Day 30 and Day 60
  Apnea-hypopnea index (AHI) is the total number of episodes of complete or partial cessation of breathing during one hour of sleep (with polysomnography or cardiorespiratory monitoring). AHI is used to assess the severity of OSAS. Calculated using the formula: (number of apnea episodes + number of hypopnea episodes) / sleep or study time.
  AHI <5 is considered the norm. Average degree of OSAS 15≤IAG <30. Severe AHI ≥30. A decrease in the indicator shows an improvement in OSAS during treatment.
The Epworth Sleepiness Scale (ESS) | Screening, Day 30 and Day 60
  The Epworth Sleepiness Scale (ESS) is a scale for measuring daytime sleepiness using a questionnaire. Helpful in diagnosing sleep disorders.
  Subjects are asked to rate the likelihood of falling asleep on a scale of increasing probability from 0 to 3 for various situations they encounter in everyday life. The scores for the eight questions are added to form a single number. A number in the range of 0-9 is considered normal, while a number in the range of 10-24 indicates that you should seek professional advice.
Pittsburgh Sleep Quality Index (PSQI) Questionnaire | Screening, Day 30 and Day 60
  The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire that assesses sleep quality over a 1 month time frame. It consists of 19 individual elements, making up 7 components that give one overall rating. Each item is weighted on a scale from 0 to 3. The overall PSQI score is then calculated by adding the scores of the seven components to give an overall score of 0 to 21, where lower scores mean healthier sleep quality.
Cardiorespiratory monitoring | Screening, Day 60
  Cardiorespiratory monitoring - is one of the main methods for diagnosing snoring and breathing disorders during sleep. It allows you to identify episodes of snoring and respiratory arrest (apnea) during sleep, to determine the level of oxygen during episodes of disturbed breathing, to reveal the relationship between apnea and disturbances in the rhythm and conduction of the heart, persistent arterial hypertension, and also to establish the degree of OSA
Native endoscopy of the upper respiratory tract with Müller's test | Screening, Day 30 and Day 60
  Upper airway endoscopy with Müller's test is performed with flexible optics in a sitting or supine position of the patient. After a forced exhalation, he inhales with his hand closed to his nose and mouth. Levels, shapes and severity of nasal, pharyngeal and laryngeal obstruction are assessed
Sleep endoscopy | Screening, Day 60
  Sleep endoscopy (drug-induced slip endoscopy (DISE)) is a research method in which the patient is immersed in a drug-induced sleep, at a certain depth of which the sound phenomenon of snoring occurs using a flexible endoscope. All parts of the nose, pharynx and larynx are examined. The degree, shape, and levels of obstruction are determined.
The intensity of pain assesment | On the day of surgery, 2 days after the surgery
  The intensity of pain is quantified using Verbal Rating Scale. The following scale of verbal assessments is applied: 0 - no pain, 1 point - mild, 2 - moderate, 3 - strong, 4 points - very strong and 5 points - unbearable pain.
Pulse oximetry | On the day of surgery, 2 days after the surgery
  Pulse oximetry is an indirect method for assessing ventilation. Estimation of the average values of saturation is important for the detection of chronic nocturnal hypoxemia and respiratory failure during sleep. A decrease in average saturation values below 90% indicates severe respiratory failure during sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Savchuk, MD, Principal Investigator — Pirogov National Medical and Surgical Center
Locations (1):
- Pirogov National Medical and Surgical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 6 months after completion of the study
Access Criteria: upon the request

REFERENCES:
- [Result] Song SA, Wei JM, Buttram J, Tolisano AM, Chang ET, Liu SY, Certal V, Camacho M. Hyoid surgery alone for obstructive sleep apnea: A systematic review and meta-analysis. Laryngoscope. 2016 Jul;126(7):1702-8. doi: 10.1002/lary.25847. Epub 2016 Jan 23. PMID 26801005
- [Result] Canzi P, Berardi A, Tinelli C, Montevecchi F, Pagella F, Vicini C, Benazzo M. Thirteen Years of Hyoid Suspension Experience in Multilevel OSAHS Surgery: The Short-Term Results of a Bicentric Study. Int J Otolaryngol. 2013;2013:263043. doi: 10.1155/2013/263043. Epub 2013 Feb 20. PMID 23509464
- [Result] Baisch A, Maurer JT, Hormann K. The effect of hyoid suspension in a multilevel surgery concept for obstructive sleep apnea. Otolaryngol Head Neck Surg. 2006 May;134(5):856-61. doi: 10.1016/j.otohns.2006.01.015. PMID 16647548